CLINICAL TRIAL: NCT05810077
Title: Feasibility of Brachial Plexus Ultrasound in Evaluation of Patients With Brachial Plexus Injuries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager Mohamed Ahmed Lotfallah, Resident, Assiut University
Other Study IDs: Brachial plexus ultrasound
Record Dates: First submitted 2023-03-16; First posted 2023-04-12 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Brachial Plexus Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of ultrasound as a diagnostic tool in assessment of patients with brachial plexus injuries before undergoing surgical exploration

DETAILED DESCRIPTION:
Ultrasound of the brachial plexus is particularly good for assessing brachial plexus injuries, nerve sheath tumors,perineural fibrosis, metastasis, some inflammatory neuropathies, neuralgic amyotrophy and post traumatic sequele

ELIGIBILITY:
Inclusion Criteria:

* all patients ages with brachial plexus injuries

Exclusion Criteria:

* patients underwent brachial plexus surgery before
* patients with surgical emphysema
* patients with serious skeletal malformations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study sample calculated using Epi . as 36 patients.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with positive ultrasound findings of brachial plexus injuries ( nerve root avulsion, nerve rupture) . | Within 2 weeks
  Number of patients with positive ultrasound findings of brachial plexus injuries ( nerve root avulsion, nerve rupture) among all patients with brachial plexus injuries then compare our results with operative findings (as the gold standard ) to estimate sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Hager M Ahmed, Master, Principal Investigator — Assist university; Nagham N Mahmood, Professor, Study Chair — Assist university